CLINICAL TRIAL: NCT00620828
Title: The Role of Intra-Operative Intracapsular Blocks in Post-Operative Pain Management Following Total Knee Arthroplasty: A Double-Blinded Randomized Controlled Trial
Brief Title: The Role of Intra-Operative Intracapsular Blocks in Post-Operative Pain Management Following Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Pro00000233; SPS# 139715
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2013-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Block Negative (Placebo Comparator): Subjects receive intra-op saline injection per protocol
  Interventions: Other: Placebo saline injection
- Block Positive (Experimental): Subjects receive intra-op Ropivicaine 0.5% injection per protocol
  Interventions: Drug: Ropivicaine 0.5%

INTERVENTIONS:
Other: Placebo saline injection — 20 cc of sterile, injectable saline
  Arms: Block Negative
Drug: Ropivicaine 0.5% — Ropivicaine
  Other Names: Hospiria
  Arms: Block Positive

SUMMARY:
The purpose of this study is to use a new combination of anesthesia techniques in an attempt to minimize early pain after surgery and improve the patient's ability to participate more fully with physical therapy. Total knee replacement patients who participate will receive the standard anesthesia. This includes a spinal nerve block as well as a femoral nerve block. The study is looking at the added benefits of including an injection of numbing medication (Bupivicaine) to the back of the knee. This injection occurs during surgery. In order to compare the outcomes we will also have a group of patients who will receive a saline injection as opposed to the numbing medication. Patients are randomly assigned to a group. Outcomes are measured up until twenty-four hours following the surgery.

DETAILED DESCRIPTION:
Research Summary

Purpose of Study This prospective, randomized, blinded controlled trial will be conducted to evaluate post-operative pain control and physical therapy outcomes in primary total knee arthroplasty (TKA) with the use of spinal analgesia and intra-operative posterior capsular injections of ropivicaine 0.5% in conjunction with a continuous femoral nerve catheter.

We believe the results of this study will show an improvement in pain control and physical therapy outcomes compared to traditional methods of analgesia in post-op total knee arthroplasty. To the best of our knowledge, there are no studies in the literature using this combination of femoral nerve analgesia and posterior capsular injection.

Certainly regional anesthesia methods such as femoral nerve blocks used alone or in conjunction with sciatic nerve blocks have improved patient pain outcome measures in total knee arthroplasty. Several studies have shown a beneficial effect of intra-articular analgesia after capsular closure. We believe our study design will combine the beneficial effects of the aforementioned methods, and ultimately improve patient pain, therapy effort, and safety through less narcotic use.

Our goal is to share these results in a peer-reviewed journal, and at national orthopaedic or anesthesia meetings. The data collected will ideally improve care and safety in the post-operative total knee arthroplasty patient.

Background and Significance Post-operative pain control in total knee arthroplasty is an area of great study in the orthopaedic surgery and anesthesia literature. The use of spinal/epidural alone or in combination with regional anesthesia is well studied in the recent literature. These techniques have significantly improved patient pain management, physical/occupational therapy outcomes, and shortened time to discharge.

Additionally, intra-articular injection of local anesthetic after capsular closure has been studied recently. Several studies have demonstrated a beneficial effect of intra-articular local anesthetic on pain outcome measures (6, 8, 9, 10, 15). Although other studies have reported more equivocal results. The impact of capsular analgesia has on post-operative pain is intriguing. Decreased afferent pain perception by the capsular nerves from local anesthetic may improve outcomes, especially in sensory distributions where regional anesthesia is inadequate or not performed.

Much study has centered on regional anesthesia, specifically the use of single shot or continuous femoral nerve blockade (4, 5, 11, 14, 16). Such studies have demonstrated a statistically significant decrease in total narcotic use, sedation scores, and visual analog pain scores. Femoral nerve blockade is now an accepted method of post-op pain control in the total knee arthroplasty patient.

Further investigation has centered on the addition of sciatic nerve blockade to femoral nerve block (1-3, 7, 12, 13). Several studies demonstrate a further improvement in pain outcomes compared to isolated femoral nerve anesthesia. Sciatic nerve blocks can slow physical therapy efforts secondary to a dense motor blockade. Equivocal results have been reported in other studies due to this motor block, however, the sensory component appears to provide improved pain outcome measures.

Femoral nerve blockade is a well-accepted modality for analgesia in total knee arthroplasty. However, femoral nerve block alone does not provide adequate anesthesia to the posterior aspect of the knee. We believe that intra-operative injection of ropivicaine 0.5% into the posterior capsule will provide analgesia analogous to the sensory component of a sciatic nerve block, while eliminating the limiting effects of the motor blockade. The combination of femoral nerve block and intra-operative posterior capsular injection will ideally yield improved pain management and physical therapy efforts above a baseline femoral nerve block.

Design and procedures This is a prospective double-blinded, randomized trial consisting of two study groups: posterior capsular saline injection (control), and the experimental posterior capsular ropivicaine 0.5% injection group. All patients will receive spinal anesthesia and a continuous femoral nerve block. Each group will include 45 patients (n = 90 patients).

All patients will have an elective primary total knee arthroplasty performed. No revision or bilateral cases will be included. Exclusion criteria will include patients with a known allergy to ropivicaine or fentanyl, a known history of narcotic abuse or chronic pain, a known diagnosis of peripheral neuropathy or complex regional pain syndrome, or a significant impediment to physical therapy participation.

Following the informed consent process, patients will receive a continuous femoral nerve block via catheter placed by experienced regional anesthesiologists at our institution. Each patient will also receive spinal anesthesia for intra-operative pain control. A standard midline skin incision with medial para-patellar arthrotomy will be performed followed by implantation of either a Next Gen (Zimmer/Warsaw, IN), or Natural Knee II (Zimmer, Warsaw, IN), or Posterior Femoral Component (PFC) Sigma (DePuy, Warsaw, IN) system. Prior to surgery, patients will be randomized to the saline or ropivicaine groups. Both groups will receive their respective injection prior to implantation of the components.

The posterior capsule of the knee will be divided in to four quadrants, each receiving a saline or ropivicaine injection per randomization. Safety measures will include standard pre-injection aspiration to check for vascular blush and intra-operative Doppler ultrasound to identify vascular structures in the posterior knee. Additionally, the anesthesiologist will not be blinded, as he/she will be responsible for assuring the appropriate medication is used, and will be closely monitoring for cardiac arrhythmias in the unlikely event that an intravascular injection occurs. Post-operatively, a standard bulky dressing will be applied. All patients will be weight bearing as tolerated post-operative day 1. A fentanyl PCA will be initiated in the PACU, and will be continued until post-operative day 2. Dosing will be calculated based on lean body mass. Continuous femoral nerve blockade will continue until post-operative day 2 as well.

Outcomes will include total PCA narcotic use, visual analog pain scale with a diagram to localize pain, and Ramsey sedation scores. This data will be collected at the following intervals: in the PACU, 4, 8, 12, and 24 hours post-operatively. We will also measure post-operative day 1 knee range of motion, total ambulation distance, and time to straight leg raise. A standard, Institutional Review Board (IRB) approved, data collection sheet will be utilized.

We hypothesize that total post-operative narcotic use, visual analog pain scores, and Ramsey sedation scores will be significantly lower in the study group (posterior capsular ropivicaine 0.5% injection). Additionally, we anticipate the knee range of motion, total ambulation distance, and time to straight leg raise to be significantly improved as well.

ELIGIBILITY:
Inclusion Criteria:

* The subject is scheduled to undergo elective total knee replacement at Duke University Hospital.
* The subject has signed the written consent form.

Exclusion Criteria:

* Known allergy to ropivacaine or hydromorphone.
* Known history of narcotic abuse or alcohol abuse.
* Known history of chronic pain.
* Known diagnosis of peripheral neuropathy or complex regional pain syndrome.
* Significant impediment to physical therapy participation.
* The surgery is a revision case.
* Patient is undergoing bilateral Total Knee Replacement.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Bolognesi, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Adult Reconstructive Surgery, Durham, North Carolina, United States

REFERENCES:
- [Background] Ben-David B, Schmalenberger K, Chelly JE. Analgesia after total knee arthroplasty: is continuous sciatic blockade needed in addition to continuous femoral blockade? Anesth Analg. 2004 Mar;98(3):747-9, table of contents. doi: 10.1213/01.ane.0000096186.89230.56. PMID 14980931
- [Background] Cook P, Stevens J, Gaudron C. Comparing the effects of femoral nerve block versus femoral and sciatic nerve block on pain and opiate consumption after total knee arthroplasty. J Arthroplasty. 2003 Aug;18(5):583-6. doi: 10.1016/s0883-5403(03)00198-0. PMID 12934209
- [Background] Davies AF, Segar EP, Murdoch J, Wright DE, Wilson IH. Epidural infusion or combined femoral and sciatic nerve blocks as perioperative analgesia for knee arthroplasty. Br J Anaesth. 2004 Sep;93(3):368-74. doi: 10.1093/bja/aeh224. Epub 2004 Jul 9. PMID 15247111
- [Background] Edwards ND, Wright EM. Continuous low-dose 3-in-1 nerve blockade for postoperative pain relief after total knee replacement. Anesth Analg. 1992 Aug;75(2):265-7. doi: 10.1213/00000539-199208000-00020. PMID 1632541
- [Background] Hirst GC, Lang SA, Dust WN, Cassidy JD, Yip RW. Femoral nerve block. Single injection versus continuous infusion for total knee arthroplasty. Reg Anesth. 1996 Jul-Aug;21(4):292-7. PMID 8837185
- [Background] Klasen JA, Opitz SA, Melzer C, Thiel A, Hempelmann G. Intraarticular, epidural, and intravenous analgesia after total knee arthroplasty. Acta Anaesthesiol Scand. 1999 Nov;43(10):1021-6. doi: 10.1034/j.1399-6576.1999.431009.x. PMID 10593465
- [Background] Lau HP, Yip KM, Jiang CC. Regional nerve block for total knee arthroplasty. J Formos Med Assoc. 1998 Jun;97(6):428-30. PMID 9650474
- [Background] Lombardi AV Jr, Berend KR, Mallory TH, Dodds KL, Adams JB. Soft tissue and intra-articular injection of bupivacaine, epinephrine, and morphine has a beneficial effect after total knee arthroplasty. Clin Orthop Relat Res. 2004 Nov;(428):125-30. doi: 10.1097/01.blo.0000147701.24029.cc. PMID 15534532
- [Background] Mauerhan DR, Campbell M, Miller JS, Mokris JG, Gregory A, Kiebzak GM. Intra-articular morphine and/or bupivacaine in the management of pain after total knee arthroplasty. J Arthroplasty. 1997 Aug;12(5):546-52. doi: 10.1016/s0883-5403(97)90178-9. PMID 9268795
- [Background] Nechleba J, Rogers V, Cortina G, Cooney T. Continuous intra-articular infusion of bupivacaine for postoperative pain following total knee arthroplasty. J Knee Surg. 2005 Jul;18(3):197-202. doi: 10.1055/s-0030-1248181. PMID 16152868
- [Background] Niskanen RO, Strandberg N. Bedside femoral block performed on the first postoperative day after unilateral total knee arthroplasty: a randomized study of 49 patients. J Knee Surg. 2005 Jul;18(3):192-6. doi: 10.1055/s-0030-1248180. PMID 16152867
- [Background] Pham Dang C, Gautheron E, Guilley J, Fernandez M, Waast D, Volteau C, Nguyen JM, Pinaud M. The value of adding sciatic block to continuous femoral block for analgesia after total knee replacement. Reg Anesth Pain Med. 2005 Mar-Apr;30(2):128-33. doi: 10.1016/j.rapm.2004.11.009. PMID 15765454
- [Background] Szczukowski MJ Jr, Hines JA, Snell JA, Sisca TS. Femoral nerve block for total knee arthroplasty patients: a method to control postoperative pain. J Arthroplasty. 2004 Sep;19(6):720-5. doi: 10.1016/j.arth.2004.02.043. PMID 15343531
- [Background] Tanaka N, Sakahashi H, Sato E, Hirose K, Ishii S. The efficacy of intra-articular analgesia after total knee arthroplasty in patients with rheumatoid arthritis and in patients with osteoarthritis. J Arthroplasty. 2001 Apr;16(3):306-11. doi: 10.1054/arth.2001.21496. PMID 11307127
- [Background] Wang H, Boctor B, Verner J. The effect of single-injection femoral nerve block on rehabilitation and length of hospital stay after total knee replacement. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):139-44. doi: 10.1053/rapm.2002.29253. PMID 11915059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 of the 79 subjects enrolled were screening failures, thus total number of subjects completing the study = 67. One patient had staged bilateral TKA so there are 66 total patients, but 67 injections given.
Pre-assignment Details: 12 of the 79 subjects enrolled were screening failures
Groups:
- Control Group: Subjects receive intra-op saline injection per protocol
- Block Group: Subjects receive intra-op Ropivicaine 0.5% injection per protocol
Period: Overall Study
Arm/Group | Control Group | Block Group
Started | 32 | 35
Number of Subjects Enrolled = 67 | 32 | 35
Completed | 32 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Block Group | Total
Number analyzed (Participants) | 32 | 35 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (2) | 66.9 (2) | 66.1 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 44
  Male | 8 | 15 | 23
Region of Enrollment [Number; unit: participants]
  United States | 32 | 35 | 67
Lean Body Weight [Mean (Standard Deviation); unit: kg] | 59.9 (12.4) | 62.9 (11.1) | 61.4 (11.75)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Score
Description: Participants were asked to rate their pain on a scale of 0 to 10 at all time intervals up to 24 hours post-injection. Scores were organized into the following categories: 3 or less (mild pain), 4 to 6 (moderate pain), 7 or higher (severe pain).
Time Frame: Post-anesthesia care unit (PACU), 4 hours, 8 hours, 12 hours and 24 hours post-injection
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Block Group: Participants received a 20 mL posterior capsular injection of ropivicaine before cementation of final components. The posterior capsule of the knee was divided into 4 quadrants, each receiving a 5 mL injection of ropivicaine.
- Control Group: Participants received a 20 mL posterior capsular injection of saline before cementation of final components. The posterior capsule of the knee was divided into 4 quadrants, each receiving a 5 mL injection of saline.
Arm/Group | Block Group | Control Group
Number analyzed (Participants) | 35 | 32
units on a scale
  PACU | 0.67 (1.4) [0 to 0] | 1.6 (2.8) [0 to 0]
  4 hours | 2.5 (2.7) | 3.6 (2.8)
  8 hours | 3.8 (2.6) | 4.9 (2.8)
  12 hours | 3.2 (1.9) | 3.9 (2.6)
  24 hours | 3.9 (2.7) | 4.9 (2.6)
Statistical Analysis 1: Comparison: Block Group vs Control Group; Patient cohort was inclusive of patient undergoing single TKA from June 2007 to July 2008. Effect size was calculated for the numeric pain rating scale at the immediate post-operative period, 4-hour, 8-hour , 12-hour, and 24-hour time periods as a means to assess post-operative pain control; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Total Fentanyl Patient-Controlled Anesthesia (PCA) Narcotic Consumption
Description: The PCA total dose at the 4-hour, 8-hour, 12-hour and 24-hour post-operative time points.
Time Frame: 4 hours to 24 hours post-op
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Block Group | Control Group
Number analyzed (Participants) | 35 | 32
micrograms
  4 hours | 22.4 (38.1) | 43.7 (71.9)
  8 hours | 95.6 (103.3) | 126.6 (106.4)
  12 hours | 173.4 (175.4) | 205.6 (177.5)
  24 hours | 418.5 (424.4) | 292.2 (402.1)
Statistical Analysis 1: Comparison: Block Group vs Control Group; Significant differences in Fentanyl PCA pump usage across study arms were assessed for the 4-8h,8-12h,and 12h-24h time frames; Test type: Superiority or Other; p = .05, ANOVA

3. Secondary Outcome: Postoperative Day 1 Physical Therapy Outcome - Ambulation Distance
Description: Ambulation distance walked by participants 24-hours post-operatively
Time Frame: 24 hours post-op
Measure: Median (Standard Deviation); unit: Feet
Arm/Group | Block Group | Control Group
Number analyzed (Participants) | 35 | 32
Feet | 38.4 (45.0) | 26.4 (27.7)
Statistical Analysis 1: Comparison: Block Group vs Control Group; This analysis was performed on data collected 24-hours post-operatively for patient cohort; Test type: Superiority or Other; p = .05, t-test, 1 sided

4. Secondary Outcome: Postoperative Day 1 Physical Therapy Outcome- Knee Extension and Flexion
Description: Knee extension and knee flexion measured at 24-hours post-operatively for patient cohort
Time Frame: 24 hours post-op
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Block Group | Control Group
Number analyzed (Participants) | 35 | 32
degrees
  Knee extension | 7.8 (4.5) | 7.0 (4.8)
  Knee flexion | 71.5 (13.9) | 69.6 (14.1)
Statistical Analysis 1: Comparison: Block Group vs Control Group; Knee extension and knee flexion measured at 24-hours post-operatively for patient cohort; Test type: Superiority or Other; p = .05, t-test, 1 sided

5. Secondary Outcome: Postoperative Day 1 Physical Therapy Outcome - Straight Leg Raise
Description: Straight Leg Raise (SLR): number of people that can perform a SLR at designated intervals
Time Frame: 4 hours, 8 hours, 12 hours and 24 hours post-op
Measure: Number; unit: participants
Arm/Group | Block Group | Control Group
Number analyzed (Participants) | 35 | 32
participants
  SLR 4 hrs | 4 | 5
  SLR 8 hrs | 13 | 5
  SLR 12 hrs | 12 | 5
  SLR 24 hrs | 13 | 6
Statistical Analysis 1: Comparison: Block Group vs Control Group; Straight leg raise data collected at 4-hours, 8-hours, 12-hours and 24-hours post-operatively for patient cohort; Test type: Superiority or Other; p = .05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Control Group | Block Group
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/35
Other Adverse Events (participants affected / at risk) | 0/32 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No